CLINICAL TRIAL: NCT04130880
Title: Reliability and Validity of the Turkish Montreal Children's Hospital Feeding Scale
Brief Title: Turkish Montreal Children's Hospital Feeding Scale
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İNAL, Principal Investigator, Hacettepe University
Other Study IDs: Turkish Montreal
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-02

CONDITIONS: Feeding Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with cerebral palsy: Children with CP who aged between 18 months and 6 years will be evaluated.
  Interventions: Diagnostic Test: Turkish Montreal Children's Hospital Feeding Scale
- Children with typical development: Children with typical development who aged between 18 months and 6 years will be evaluated.
  Interventions: Diagnostic Test: Turkish Montreal Children's Hospital Feeding Scale

INTERVENTIONS:
Diagnostic Test: Turkish Montreal Children's Hospital Feeding Scale — The Turkish version of the Montreal Children's Hospital Feeding Scale, and the Behavioral Pediatrics Feeding Assessment Scale will be completed.

SUMMARY:
The purpose of this study is to test the reliability and validity of the Turkish Montreal Children's Hospital Feeding Scale.

DETAILED DESCRIPTION:
The purpose of this study is to test the reliability and validity of the Turkish Montreal Children's Hospital Feeding Scale. The internal consistency, test-retest reliability, and criterion validity of Turkish Montreal Children's Hospital Feeding Scale will be investigated. The internal consistency will be assessed using Cronbach's alpha. Intraclass correlation coefficient (ICC) value with 95 % confidence intervals will be calculated for test-retest reliability. The criterion validity of the scale will be determined by assessing the correlation between the Turkish Montreal Children's Hospital Feeding Scale and Behavioral Pediatrics Feeding Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy
* Children with typical development
* Aged between 18 months- 6 years

Exclusion Criteria:

* Who aged under the age of 18 months and above the age of 6 years.

Ages: 18 Months to 6 Years | Sex: All
Age Groups: Child
Study Population: Children with cerebral palsy and Children with typical development
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Montreal Children's Hospital Feeding Scale | 2 months
  The Montreal Children's Hospital Feeding Scale is used to evaluate feeding disorders. It has 14 items which are scored on a 7 point Likert scale. Seven items are scored from the negative to positive direction, and the other seven from the positive to negative direction. The primary feeder marks each item according to frequency or difficulty level of a particular behaviour or the level of parental concern. The total feeding problem score is obtained by adding the scores for each item after reversing the scores of seven items from negative to positive.

SECONDARY OUTCOMES:
Behavioral Pediatrics Feeding Assessment Scale | 2 months
  The Behavioral Pediatrics Feeding Assessment Scale is a widely used parent-report measure of mealtime and feeding behavior. It has 35 items.Greater overall scores indicate higher levels of problematic mealtime and feeding behavior.

CONTACTS AND LOCATIONS:
Overall Officials: ÖZGÜ İNAL, Principal Investigator — Trakya University
Locations (1):
- Özgü İnal, Edirne, Turkey (Türkiye)